CLINICAL TRIAL: NCT06132022
Title: The Effect of Mandala Application on Anxiety Level and Caregiver Burden in Palliative Caregivers: A Randomized Controlled Trial
Brief Title: The Effect of Mandala Application on Anxiety Level and Caregiver Burden in Palliative Care
Acronym: MANDALAPLİC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bartın Unıversity (Other)
Responsible Party: Principal Investigator, Necmiye ÇÖMLEKÇİ, Principal Investigator, Bartın Unıversity
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 27042
Record Dates: First submitted 2023-05-30; First posted 2023-11-15 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Palliative Care; Caregiver; Anxiety; Mandala; Caregiver Burden
MeSH Terms: conditions — Anxiety Disorders; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: Rondomized Controlled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will be asked to practice the mandala twice a week, for 30 minutes, for a month. At the end of one month, the scales will be applied again.
  Interventions: Other: Mandala
- Control group (Placebo Comparator): Caregivers in the control group will not take any action, and at the end of one month, after the scales have been applied, they will be offered mandala applications.
  Interventions: Other: Routine care

INTERVENTIONS:
Other: Mandala — Mandala work is one of the non-pharmacological approaches and is used to support patients and caregivers in various diseases. Mandala is a method that anyone can apply based on coloring a circular shape.
  Arms: Intervention group
Other: Routine care — The clinic's routine information will be given to the caregivers of the control group.
  Arms: Control group

SUMMARY:
The caregivers of palliative care patients can also be negatively affected during the palliative care process. Especially family caregivers may experience difficulties in physical, social, economic, and psychological aspects. Non-pharmacological approaches are utilized to cope with these difficulties. The mandala study is one of the non-pharmacological approaches and has been utilized to support patients and caregivers in various illnesses. Mandala is a method that anyone can apply, based on coloring circular patterns. Recent studies have reported that mandala contributes to improving psychological and physiological well-being. This study is designed in a randomized controlled design to examine the effects of mandala application on anxiety levels and caregiver burden in palliative care caregivers. Caregivers who meet the inclusion and exclusion criteria will be randomly assigned to two groups using a computer program. Both groups of caregivers will be administered an information form, the STAI XT-1 State-Trait Anxiety Inventory, and the Zarit Burden Interview Scale. Then, the intervention group will be asked to apply mandala twice a week for 30 minutes for one month. After one month, the scales will be administered again. The caregivers in the control group will not receive any intervention, and after one month, the scales will be administered, and mandala application will be suggested. According to G Power analysis, with a Type I error (α) of 0.05 and a power (1-β) of 0.80, the minimum sample size that will meet the requirements is determined to be a total of 86 individuals (experimental: 43, control: 43). Considering potential sample loss, the aim is to reach 45 participants in each group. The statistical analysis of the data will be performed using SPSS version 22.0. Descriptive statistics such as frequency, median, standard deviation, mean, minimum, maximum, percentage, Kolmogorov-Smirnov test for normal distribution (N>30), skewness, and kurtosis will be used for sociodemographic characteristics. Correlation tests will be used for scale relationships, and ANOVA, Kruskal-Wallis, t-test, or Mann-Whitney U test and post-hoc tests will be used for scale comparisons according to independent variables. The significance level will be accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* have reached the age of 18
* Willingness to participate in the study
* Being able to read and write
* Having no problems in verbal communication
* Providing free care

Exclusion Criteria:

* Providing paid care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
STAI XT-1 State-Trait Anxiety Scale | 4 weeks
  score anxiety: While the state anxiety scale shows the level of anxiety in a certain situation, the trait anxiety scale evaluates the level of anxiety experienced by the individual regardless of the situation. Scores on both scales range between 20 and 80. High scores indicate high anxiety level, low scores indicate low anxiety level.
Zarit Care Burden Scale | 4 weeks
  Care Burden Scale: The scale, which can be completed by asking the caregivers themselves or the researcher, consists of 22 statements that determine the impact of caregiving on the individual's life. With this, the caregiver/patient relationship, the caregiver's health status, psychological comfort, social life and economic burden can be evaluated. The evaluation of scale, in which all items are clearly stated, is made on the basis of the total score. As the score increases, the burden of care also increases and a maximum score of 88 is obtained from the scale. Points obtained; It was evaluated by grading as (0-20) little/no burden, (21-40) moderate burden, (41-60) severe burden and (61-88) extreme burden.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Atlas University, Istanbul, Kağıthane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data will be stored in flash memory and shared with other researchers when necessary.